CLINICAL TRIAL: NCT06723795
Title: Early Cardiovascular Risk Assessment of Patients With COPD During Respiratory Exacerbation for the Identification and Treatment of Cardiovascular Comorbidity
Brief Title: Cardiovascular Assessment and Treatment During COPD Exacerbation to Improve Diagnosis and Outcomes
Acronym: CATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 0510-24-TLV
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Cardiovascular Diseases
Keywords: COPD exacerbation; Cardiovascular disease; Comorbidity; Diagnosis; Screening
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases; Disease

STUDY DESIGN:
Intervention Model Description: Given the unique intervention, it is expected that the department's daily practices may change during the study due to exposure to the intervention (increased cardiovascular screening and treatment in COPD patients). This could directly impact the intervention's effectiveness. In addition, the quality of treatment and personnel in each department might affect the compliance with the cardiologists recommendations. Therefore, randomization will not be made at the individual or department level, but rather consecutive patients will first be recruited to the control group, followed by 3 weeks of wash-out, and then recruited for the intervention.
  COPD patients will be identified by their treating physicians and referred to the research team.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The interviewer in the 1, 3, 6 and 12 months phone call follow-up will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients will be evaluated by a pulmonologist during their admission, in addition to a cardiologist, aiming to identify cardiovascular comorbidities including dyslipidemia, diabetes, hypertension, ischemic heart disease, heart failure, valvular disease, personal or family history of ischemic heart disease, and smoking. Part of the evaluation will include assessing the management of diagnosed cardiovascular conditions. Finally, recommendations for further investigation or initiation of drug treatment will be made.
  Interventions: Other: Cardiologist evaluation; Other: Pulmonologist evaluation
- Control (Active Comparator): Patients will be evaluated by a pulmonologist during their hospitalization, who will focus on their pulmonary condition, optimize basic treatment, and recommend continued follow-up as needed.
  Interventions: Other: Pulmonologist evaluation

INTERVENTIONS:
Other: Cardiologist evaluation — The cardiology consultation will include the following: a structured interview (see Appendix A), physical examination, review of laboratory tests including HbA1c, lipid profile, BNP, ECG, and POCUS (point-of-care ultrasound) to assess heart contraction and valve function.
  Arms: Intervention
Other: Pulmonologist evaluation — optimize basic treatment, and recommend continued follow-up as needed.

SUMMARY:
This is a research study involving patients hospitalized for COPD flare-ups. Patients will be randomly assigned to two groups: one group will only see a pulmonologist (lung doctor), and the other group will also be seen by a cardiologist (heart doctor) during their hospital stay. Both groups will fill out a questionnaire, and the pulmonologist will review their lung disease, adjust their treatment, and recommend follow-up care. The cardiologist will also assess the second group for heart diseases (like high cholesterol, diabetes, heart disease, high blood pressure, or heart failure) and start or adjust heart treatment if needed. Both groups will be followed up by phone 1, 3, 6 and 12 months later to check for changes in treatment, new heart problems, COPD flare-ups, or death.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized study involving patients hospitalized for COPD exacerbation. Eligible patients will be identified either by the internal medicine department doctors or by reviewing the admission diagnoses of hospitalized patients in the hospital's database. After obtaining informed consent, the patients will be randomized into two groups.

Both groups will complete a background questionnaire and will be assessed by a pulmonologist during the hospitalization, who will focus on their lung disease, optimize basic treatment, and recommend follow-up as needed. The intervention group will undergo an additional evaluation by a cardiologist during the hospitalization, who will check for cardiovascular diseases (such as hyperlipidemia, diabetes, ischemic heart disease, hypertension, or heart failure) and adjust or start treatment according to new or existing diagnoses.

Both groups will receive follow-up phone calls about 1, 3, 6, and 12 months later to evaluate any changes in treatment following the intervention, new diagnoses or events of cardiovascular diseases, COPD exacerbations, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Documented COPD (based on lung function tests, symptoms and relevant treatment).
* Aged 18-75 years.
* Mentally competent to understand and follow medical recommendations.

Exclusion Criteria:

* Under 18 years of age.
* Unable to provide consent.
* Unstable concurrent disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular-related treatment change in 6 months | From enrollment to 6 months follow-up call
  New pharmacological treatment or intervention (e.g., angiography, surgery) for cardiovascular disease, including diabetes, hypertension, dyslipidemia, ischemic heart disease, stroke, valvular disease, or heart failure compared to at inclusion.

SECONDARY OUTCOMES:
Diagnosis of new cardiovascular comorbidity | From inclusion to hospital discharge
  Identification of new cardiovascular comorbidities, including diabetes, dyslipidemia, ischemic heart disease, valvular disease, or heart failure.
Extended diagnosis of new cardiovascular comorbidity | At 6 months after enrollment.
  Identification of new cardiovascular comorbidities, including diabetes, dyslipidemia, ischemic heart disease, valvular disease, or heart failure.
Adverse outcomes | At 3 and 6 months from study enrollment
  Combined outcome of Major Adverse Cardiovascular Events (MACE - stroke, myocardial infarction, cardiovascular mortality) and readmissions or mortality due to COPD
MACE | At 3 and 6 months from enrollment
  Occurrence of MACE - MACE - stroke, myocardial infarction, cardiovascular mortality.
Time to MACE | 6 months from enrollment
  Time from enrollment to first MACE - stroke, myocardial infarction, cardiovascular mortality
COPD exacerbations | 3 and 6 months from enrollment
  Amount of COPD exacerbations, defined as an event characterized by an acute change in the patient's baseline dyspnoea, cough, and/or sputum that warrant a change in regular medication.
COPD severe exacerbations | 6 months from study recruitment
  Amount of COPD exacerbations that leads to hospitalization

OTHER OUTCOMES:
Time to COPD exacerbation | 6 moths from enrollment
  Time to COPD exacerbation, defined as an event characterized by an acute change in the patient's baseline dyspnea, cough, and/or sputum that warrant a change in regular medication.
Adherence to new treatment | 6 months from enrollment
  Adherence to newly initiated pharmacological treatment from the study intervention
Smoking cessation | 6 and 3 months from enrollment
  Rates of smoking cessation between the intervention and control groups among smokers
Specialists follow-up | 6 months from enrollment
  Rate of patients with cardiologist and pulmonologist visits
Post-Hoc analysis - Treatment | 12 months from recruitment
  New pharmacological treatment or intervention (e.g., angiography, surgery) for cardiovascular disease, including diabetes, hypertension, dyslipidemia, ischemic heart disease, stroke, valvular disease, or heart failure compared to at inclusion.
Post-HOC analysis - diagnoses | 12 months from recruitment
  Identification of new cardiovascular comorbidities, including diabetes, dyslipidemia, ischemic heart disease, valvular disease, or heart failure.
Post-HOC analysis - COPD exacerbations | 12 months from recruitment
  COPD exacerbations requiring steroids or hospital arrival
Post-HOC analysis - MACE | 12 months from recruitment
  Occurance of MACE between the intervention and control

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not permitted as per our institution review board.

REFERENCES:
- [Background] Vogelmeier C, Simons S, Garbe E, et al. Increased risk of severe cardiovascular events following exacerbations of COPD: a multi-database cohort study. Eur Respir J. 2023;62(suppl 67). doi:10.1183/13993003.congress-2023.PA3013
- [Background] Swart KMA, Baak BN, Lemmens L, Penning-van Beest FJA, Bengtsson C, Lobier M, Hoti F, Vojinovic D, van Burk L, Rhodes K, Garbe E, Herings RMC, Nordon C, Simons SO. Risk of cardiovascular events after an exacerbation of chronic obstructive pulmonary disease: results from the EXACOS-CV cohort study using the PHARMO Data Network in the Netherlands. Respir Res. 2023 Nov 21;24(1):293. doi: 10.1186/s12931-023-02601-4. PMID 37990197
- [Background] Hawkins NM, Peterson S, Ezzat AM, Vijh R, Virani SA, Gibb A, Mancini GBJ, Wong ST. Control of Cardiovascular Risk Factors in Patients with Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2022 Jul;19(7):1102-1111. doi: 10.1513/AnnalsATS.202104-463OC. PMID 35007497
- [Background] Feary JR, Rodrigues LC, Smith CJ, Hubbard RB, Gibson JE. Prevalence of major comorbidities in subjects with COPD and incidence of myocardial infarction and stroke: a comprehensive analysis using data from primary care. Thorax. 2010 Nov;65(11):956-62. doi: 10.1136/thx.2009.128082. Epub 2010 Sep 25. PMID 20871122